CLINICAL TRIAL: NCT02617134
Title: Immunotherapy With Chimeric Antigen Receptor-Modified T Cells for MUC1 Positive Advanced Refractory Solid Tumor
Brief Title: CAR-T Cell Immunotherapy in MUC1 Positive Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-021-002
Record Dates: First submitted 2015-11-26; First posted 2015-11-30 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-07

CONDITIONS: Malignant Glioma of Brain; Colorectal Carcinoma; Gastric Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-T cell immunotherapy (Experimental): Enrolled patients will receive CAR-T cell immunotherapy with a novel specific chimeric antigen receptor targeting MUC1 antigen by infusion.
  Interventions: Biological: anti-MUC1 CAR-T cells

INTERVENTIONS:
Biological: anti-MUC1 CAR-T cells
  Other Names: anti-MUC1-CAR transduced autologous T cells

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-T cell immunotherapy in patients with MUC1 positive relapsed or refractory solid tumor.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with MUC1+ malignancies in patients with no available curative treatment options who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled:

* Eligible diseases: MUC1+ malignant glioma of brain, colorectal carcinoma and gastric carcinoma.

  1a. Malignant Glioma of Brain Failure after previous standard of care initial treatment of glioblastoma multiforme; documentation by magnetic resonance imaging (MRI) of an interval increase in nodular gadolinium enhancement consistent with recurrent malignant glioma suitable for therapeutic re-resection; previous pathological diagnosis of World Health Organization (WHO) Grade IV glioma;

  1b. Colorectal Carcinoma Patients must have histologically proven adenocarcinoma primary to the colon or rectum and clinical or pathologic evidence of distant metastasis;

  1c. Gastric Carcinoma Histologically confirmed adenocarcinoma of the stomach, gastroesophageal junction or esophagus; metastatic disease or locally advanced disease not amenable to curative surgery.
* Patients 18 years of age or older, and must have a life expectancy > 12 weeks.
* MUC1 is expressed in malignancy tissues by immuno-histochemical (IHC).
* Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
* Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
* Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR T cells.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
* Ability to give informed consent.

Exclusion Criteria:

* The transduction efficiency of the T cells is less than 30% or the amplification of the T cells via artificial antigen presenting cell (aAPC) stimulation is less than 5 times.
* Pregnant or nursing women may not participate.
* Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
* History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products.
* The existence of unstable or active ulcers or gastrointestinal bleeding.
* Patients with portal vein vascular invasion or extrahepatic, are excluded from this study.
* Patients with a history of organ transplantation or are waiting for organ transplantation.
* Patients need anticoagulant therapy (such as warfarin or heparin).
* Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).
* Patients treated by radiotherapy within 4 weeks prior the first apheresis.
* Patients using fludarabine or cladribine chemotherapy within two years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Adverse events attributed to the administration of the anti-MUC1 CAR-T cells | 2 years
  Determine the toxicity profile of the MUC1 targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Objective Response Rate | Safety follow-up is 100 days from last CAR-T infusion.
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Ph.D., Principal Investigator — PersonGen BioTherapeutics (Suzhou) Co., Ltd.
Locations (1):
- PersonGen Biomedicine (Suzhou) Co., Ltd., Suzhou, Jiangsu, China